CLINICAL TRIAL: NCT05302375
Title: Developing and Testing an Online Pathway From Screening to Treatment for Depression in Oncology: iPath*D (Aim 2)
Acronym: iPath Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul J. Barr, Associate Professor, Trustees of Dartmouth College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY02002016; R21CA249767 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Depression
Keywords: shared decision making; decision aid; depression
MeSH Terms: conditions — Neoplasms; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iPath*D (Experimental): An online platform that connects patients screening positive for clinically significant depression in cancer settings to a range of online and inperson evidence-based treatments, facilitated by an interactive DA.
  Interventions: Other: iPath*D

INTERVENTIONS:
Other: iPath*D — Online pathway from screening to treatment for depression in cancer patients.

SUMMARY:
The purpose of this study is to determine the extent to which an online pathway to depression treatment (iPath*D) is acceptable and usable to patients receiving cancer treatment who report symptoms of depression.

DETAILED DESCRIPTION:
The investigators will determine the extent to which an online pathway to depression treatment (iPath*D) is acceptable and usable to patients receiving cancer treatment who report symptoms of depression. iPath*D will be designed to increase screening, mental health literacy, and treatment access. Patients will access their iPath*D account online to review their PHQ-9 score and its interpretation, followed by an interactive depression decision aid comparing information on a range of online and in-person treatment options. Upon review of the decision aid, participants will be able to directly connect to a treatment path via embedded hyperlinks in the decision aid.

The investigators will determine the usability, acceptability, and feasibility of iPath*D. The investigators will explore the hypothesis that iPath*D will be highly usable, acceptable to patients, feasible to implement, and will result in improved mental health literacy, and greater treatment access. The tool for the study was developed during a preliminary portion (Aim 1) of the project, under D-H IRB number STUDY02001240 .

This approach uses an open-label, single arm pilot, with adult patients receiving treatment for cancer in a rural cancer clinic, St Johnsbury, VT (Dartmouth Cancer Center North) (n=30) with moderate-severe depression, Aim 2 of the project.

ELIGIBILITY:
Inclusion criteria

1. Adults (≥18 years)
2. New patients who are beginning treatment at Dartmouth Cancer Center North and returning for their chemo teach or radiation simulation visit
3. Can communicate in English
4. PHQ-9 ≥10 and ≤27

Exclusion criteria

1. Mild Depression (PHQ-9 ≥10)
2. Individuals who screen positive for suicidal ideation with method, intent, plan or a recent prior suicide/self-harm attempt, as determined by a positive endorsement of items 3, 4, 5 or 6 on the Columbia-Suicide Severity Rating Scale (C-SSR).
3. Individuals with bipolar disorder or psychosis (documented in the EMR)
4. Individuals currently receiving treatment for a mental health condition (documented in the EMR or self-reported during eligibility screening)
5. Significant cognitive impairment (Callahan's Six Item Screener of cognitive function ≤ 4; Self-reported during eligibility screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
System usability | 2 weeks
  System Usability Scale (10 items; mean ≥68/100),
Acceptability of intervention | 2 weeks
  Acceptability of Intervention Measure (4 items), mean ≥4/5
Feasibility of intervention | 2 weeks
  Feasibility of Intervention Measure (4 items), mean ≥4/5
Change in number of patients selecting a treatment path to access | 2 weeks, 4 weeks, 6 weeks
  Click on link to access online treatment service | indicate in self-report survey accessing local resources
Change in Mental Health Literacy (MHL) | Baseline, 2 weeks
  A modified 10-item version for the validated multiple choice questionnaire (MCQ) for depression assesses treatment knowledge, understanding & beliefs. Higher scores indicate higher MHL.

SECONDARY OUTCOMES:
Change in PHQ-9 completion (exploratory outcome) | Baseline, 2 weeks, 4 weeks, 6 weeks
  Number of patients who complete Patient Health Questionnaire (PHQ-9), a validated nine item depression scale. A score total of 0-4 points equals "normal" or minimal depression. Scoring between 5-9 points indicates mild depression, 10-14 points indicates moderate depression, 15-19 points indicates moderately severe depression, and 20 or more points indicates severe depression.
Change in treatment initiation (exploratory outcome) | 2 weeks, 4 weeks, 6 weeks
  Proportion of patients who self-report treatment initiation e.g., fill antidepressant prescription, visited with psychiatrist for talk therapy, began a cCBT program, or other service
Change in treatment adherence (exploratory outcome) | 2 weeks, 4 weeks, 6 weeks
  Proportion of patients who self-report continued adherence to treatment e.g., antidepressant refill (yes/no), number of talk therapy sessions completed, or Computerised Cognitive Behavioural Therapy (cCBT) modules completed
Decisional regret (exploratory outcome) | 6 weeks
  The Decisional Regret Scale assesses satisfaction with a healthcare decision (5-items, scores range from 0-100, with higher scores indicating high regret)
Change in PHQ-9 score (exploratory outcome) | Baseline, 2 weeks, 4 weeks, 6 weeks
  Response; 5-point reduction in baseline PHQ-9 score. Remission; PHQ-9 score of <5 points
Change in quality of life (exploratory outcome) | Baseline, 6 weeks
  Functional Assessment of Cancer Therapy-General (FACT-G) scale (27-items, scores range from 0-108 with higher scores indicating higher quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Barr, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth Cancer Center St. Johnsbury, Saint Johnsbury, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of this study, the investigators plan to make available, upon request, a public use file of all participant-level study data. Investigators will use appropriate de-identification and security measures. Plain-language descriptions of data sharing plans will be included in informed consents.
  Dartmouth College will retain ownership and all rights to all intellectual property and will provide public access to data. Appropriate documentation will also be provided regarding information about the methodology and procedures used to collect the data, details about codes and definitions of variables.
Time Frame: At the time of publication or at the end of the grant period, whichever comes first.
Access Criteria: De-identified data will be available upon request from the PI to qualified investigators, with appropriate IRB approval, and for research purposes only.